CLINICAL TRIAL: NCT05590013
Title: Determining to the Effect of Pectointercostal and ESP Block on Postoperative Analgesia During Open Heart Surgery
Brief Title: Effect of Pectointercostal+ESP Block on Postoperatif Analgesia in Open Heart Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, ebru biricik, Associate Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pectointercostal and ESP block
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2022-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pectointercostal and ESP (Active Comparator): Ultrasound (USG) guided erector spinae block will perform at T6 level (bilaterally) and pectointercostal plane block at 4-5 intercostal space to the 30 patients under general anaesthesia in Group block . Sevoflurane+remifentanil and O2/air combination will perform to the all patients during the surgery. Totally bupivacaine %0.25 2.5 mg/kg will use for blocks and 1 ml epinephrin will add to the each local anesthetic solutions in each side.10 ml %0.25 bupivacain will apply to the chest tube area at the end of surgery.
  Interventions: Drug: Pectointercostal and ESP block
- Control Group (Placebo Comparator): Block will not perform to the control group.
  Interventions: Drug: Pectointercostal and ESP block

INTERVENTIONS:
Drug: Pectointercostal and ESP block — Pectointercostal plane block will apply at the 4-5. intercostal space and ESP block will apply athe T6 level bilaterally
  Other Names: Fascial plane blocks

SUMMARY:
American Society of Anaesthesiologist physical status II-III, aged between 18-65, 60 patients which underwent open cardiac surgery will recruited to this study. These subjects will Ultrasound (USG) guided erector spinae block will perform at T6 level (bilaterally) and pectointercostal plane block at 4-5 intercostal space to the all patient under general anaesthesia. Totally bupivacaine %0.25 2.5 mg/kg will use blocks and 1 ml epinephrin will add to the each local anesthetic solutions. 10 ml %0.25 bupivacain will apply to the chest tube area at the end of surgery. 0.1 microgram/kg morphine will apply intravenously at last 30 minutes of surgery postoperative analgesia to all patients. Postoperative pain assessment will perform with visual analog scale (VAS)

DETAILED DESCRIPTION:
American Society of Anaesthesiologist physical status II-III, aged between 18-65, 60 patients which underwent open cardiac surgery will recruited to this study. The patients were randomly allocated into two groups (1:1), via a computer-generated randomization list. Ultrasound (USG) guided erector spinae block will perform at T6 level (bilaterally) and pectointercostal plane block at 4-5 intercostal space to the 30 patients under general anaesthesia in Group block and block will not perform to the control group. Sevoflurane+remifentanil and O2/air combination will perform to the all patients during the surgery. Totally bupivacaine %0.25 2.5 mg/kg will use for blocks and 1 ml epinephrin will add to the each local anesthetic solutions in each side.10 ml %0.25 bupivacain will apply to the chest tube area at the end of surgery. 0.1 microgram/kg morphine intravenously will apply for postoperative analgesia to the all patients at last 30 minutes of surgery. Postoperative pain assessment will perform with visual analog scale (VAS). VAS, morphine consumption and complications will record.Paracetamol 10 mg/kg will repeat to the all patients at the 12th of postoperative period, intravenously. The patient controlled anesthesia with morphin will apply to the all patients. If the VAS score is higher than 4, the rescue analgesic diclofenac Na 75 mg will administer intravenously.

ELIGIBILITY:
Inclusion Criteria:

* ASA II-III patients
* The patients who will operate for open heart surgery

Exclusion Criteria:

* The patients with Coagulopaty
* Allergy with local anesthetics
* infection at the injection sites
* Obesity (BMI >35kg/m2)
* Liver and/or kidney failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative analgesia | 24 hours in Postanesthesia care unit (PACU)
  Visual analog scale (VAS) scores at the postoperative 24th hours. VAS scores define pain scores between 0-10. 0 reflects nopain, 10 reflects the worst pain.
Morphine consumption | 24 hours in Postanesthesia care unit (PACU)
  Postoperative morphine consumption during the postoperative 24th hours

SECONDARY OUTCOMES:
Ekstübation time | First 6 hours at Postanesthesia care unit (PACU)
  Time between end of the surgery and extubation of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Biricik, Study Chair — Cukurova University
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No